CLINICAL TRIAL: NCT06694714
Title: Characterizing and Comparing the Duration of Local Anesthetic in Dermatologic Surgery - Fourth Arm
Brief Title: Split Face Study of the Duration of Local Anesthetics - Fourth Arm
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-10025244-1
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Two volumes of local anesthetic will be injected into the nasal skin of each participant by a dermatologic surgeon (PI of the study, Dr. Kira Minkis, KM). Dr. Minkis will be unblinded to the laterality of the anesthetic volumes and will not be involved in further assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.5 ml Lidocaine with epinephrine vs. 1.0 ml Lidocaine with epinephrine (Experimental): Each side of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed. Participants in this arm will receive an injection of 0.5ml of Xylocaine + epinephrine 1:100,000 (lidocaine + epinephrine 1:100,000), buffered 1/10 with sodium bicarb into one side of the nose (nasal ala) and 1.0 ml of Xylocaine + epinephrine 1:100,000 (lidocaine + epinephrine 1:100,000), buffered 1/10 with sodium bicarb into the opposite nasal ala. Laterality of each anesthetic volume administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes on both sides of the face, until the patient reports return of a sharp sensation upon the pinprick test.
  Interventions: Drug: 0.5 ml lidocaine + epinephrine 1:100,000; Drug: 1.0 ml lidocaine + epinephrine 1:100,000
- 1.0 ml Lidocaine with epinephrine vs 0.5 ml Lidocaine with epinephrine (Experimental): Each side of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed. Participants in this arm will receive an injection of 1.0ml of Xylocaine + epinephrine 1:100,000 (lidocaine + epinephrine 1:100,000), buffered 1/10 with sodium bicarb into one side of the nose (nasal ala) and 0.5 ml of Xylocaine + epinephrine 1:100,000 (lidocaine + epinephrine 1:100,000), buffered 1/10 with sodium bicarb into the opposite nasal ala. Laterality of each anesthetic volume administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes on both sides of the face, until the patient reports return of a sharp sensation upon the pinprick test.
  Interventions: Drug: 0.5 ml lidocaine + epinephrine 1:100,000; Drug: 1.0 ml lidocaine + epinephrine 1:100,000

INTERVENTIONS:
Drug: 0.5 ml lidocaine + epinephrine 1:100,000 — 0.5 ml lidocaine + epinephrine 1:100,000, buffered 1/10 with sodium bicarb
Drug: 1.0 ml lidocaine + epinephrine 1:100,000 — 1.0 ml lidocaine + epinephrine 1:100,000, buffered 1/10 with sodium bicarb

SUMMARY:
This is a research study to compare how long injectable pain medications (anesthetics) commonly used in dermatologic surgery are effective for. The investigators will investigate the role of anesthetic volume on the duration of action at highly vascular sites.

DETAILED DESCRIPTION:
The investigators seek to further investigate how the vascularity of an anatomical region influences the duration of local anesthetics during dermatologic surgery. The investigators hypothesize that regional vascularity, by increasing the rate of uptake and removal of the anesthetic from the infiltrated site, will significantly reduce the duration of action of increased doses of infiltrative anesthesia. Specifically, the investigators will compare the duration of a commonly used local anesthetic (lidocaine ± epinephrine) injected at two different volumes at the nasal ala. The investigators will use a modification of a previously published approach of non-invasive pinprick testing to assess the duration of local anesthesia. The investigators aim to demonstrate that there will be no clinically significant difference in the duration of action of varying volumes of the same local anesthetic injected at bilateral areas of the face.

This study record uses the same protocol document of a previous study under Clinical Trials record NCT05767749, but documents a fourth arm for which data will be analyzed separately from data in NCT05767749

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Normal skin sensation at both nasal ala assessed by pinprick
* Ability to provide informed consent

Exclusion Criteria:

* Previous adverse reaction to local anesthetic or any components of the local anesthetics being evaluated
* Pregnant or breastfeeding volunteers (assessed by self-report)
* Patients taking monoamineoxidase inhibitors (MAOI) or antidepressants of the triptyline or imipramine types

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to Return to Baseline Sensation, as Determined by Binary Outcomes (Yes/no) in 15 Minute Increments | Up to 4 hours.
  To determine whether the time to return to baseline sensation differs significantly between each pair of anesthetics, the investigators will measure the time to return to baseline sensation at each anesthetized site by asking participants at 15 minute intervals if they can feel a sharp sensation at the site. Sterile needles will be used. The return of the sensitivity will be determined using binary outcomes (yes/no) and recorded on a standardized template. The maximum difference in anesthetic duration that the investigators consider "not different" from a clinical standpoint is 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Kira Minkis, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No